CLINICAL TRIAL: NCT06783114
Title: A Clinical Study to Evaluate the Efficacy and Safety of Recombinant Botulinum Toxin Type A (YY001) for Injection in The Treatment of Upper Limb Spasticity in Adults (REHAB-1)
Brief Title: A Clinical Study on Recombinant Botulinum Toxin Type A (YY001) for Injection in The Treatment of Upper Limb Spasticity in Adults
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chongqing Claruvis Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YY001-002-CN01
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Spasticity
Keywords: YY001; Recombinant Botulinum Toxin Type A; Botulinum Toxin; Upper limb spasticity
MeSH Terms: interventions — Injections; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Placebo- and active-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): Single injection with Recombinant Botulinum Toxin Type A for injection (YY001) in upper limb spasticity
  Interventions: Biological: Recombinant Botulinum Toxin Type A for injection (YY001)
- Active-Controlled Group (Active Comparator): Single injection with BOTOX® in upper limb spasticity
  Interventions: Biological: BOTOX®
- Placebo-Controlled Group (Placebo Comparator): Single injection with placebo in upper limb spasticity
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant Botulinum Toxin Type A for injection (YY001) — Single treatment, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), intramuscular injection, the total injection dose is 200-400 U.
  Arms: Treatment Group
Biological: BOTOX® — Single treatment, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), intramuscular injection, the total injection dose is 200 U.
  Arms: Active-Controlled Group
Biological: Placebo — Single treatment, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), intramuscular injection.
  Arms: Placebo-Controlled Group

SUMMARY:
This is a randomized, double-blind, multi-center phase II/III study to evaluate the efficacy and safety of Recombinant Botulinum Toxin Type A (YY001) for injection in the treatment of upper limb spasticity in adults

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old inclusive, at the time of signing the informed consent, regardless of gender.
2. Subjects with unilateral hemiplegia due to stroke (with a time interval of ≥ 3 months from stroke onset to randomized enrollment) exhibiting upper limb spasticity.
3. Subjects with Disability Assessment Scale score of at least 2 on the Principal Target of Treatment (one of four functional domains: hygiene, dressing, limb position and pain).
4. If taking oral antispasticity, the dosage must be stable for at least 1 month prior to randomized enrollment.
5. If the study limb receives physical therapy or occupational therapy, the frequency, type, and intensity must be stable for at least 3 weeks prior to randomized enrollment.

Exclusion Criteria:

1. History of allergy to any component of the experimental drugs.
2. Previous use of any botulinum toxin within 6 months prior to randomized enrollment, or plan to use other botulinum toxins not specified in the study protocol during the study.
3. Fixed contractures of the studied limb.
4. Any medical condition that may increase the risk to the subject when using Botulinum Toxin Type A.
5. Need for treatment with drugs that interfere with neuromuscular function during the study.
6. Plan or anticipate to use new antispasticity drugs during the study.
7. History of epilepsy.
8. Pregnant or breastfeeding women.
9. Participation in other drug/device clinical trials within 1 month prior to randomized enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Modified Ashworth Scale (MAS) Score of Primary Target Clinical Pattern at Week 4 | Week 4 after treatment
  Primary target clinical pattern was defined by investigator for each subject at baseline visit and was either flexed elbow or flexed wrist or clenched fist.
  The Modified Ashworth Scale is well known and commonly used in clinical trials with spasticity. It was used to categorize severity of spasticity by judging resistance to passive movement. It is a 6-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA) Score at Week 1, Week 4, Week 8 and Week 12 | Week 1, Week 4, Week 8 and Week 12 after treatment
  The Physician's Global Assessment is used to measure the investigator's impression of change due to treatment. The response option is a common 7-point scale that ranges from -3 = very much worse to +3 = very much improved.
Change From Baseline in MAS Score of Primary Target Clinical Pattern at Week 1, Week 8, Week 12 | Week 1, Week 8 and Week 12 after treatment
Response Rates on MAS Calculated for the Primary Target Clinical Pattern at Week 1, Week 4, Week 8 and Week 12 | Week 1, Week 4, Week 8 and Week 12 after treatment
  Primary target clinical pattern was defined by investigator for each subject at baseline visit and was either flexed elbow or flexed wrist or clenched fist.
  Subjects with a MAS reduction of one point were defined as responder.
Changes From Baseline in Disability Assessment Scale (DAS)- Principal Therapeutic Target Domain at Week 1, Week 4, Week 8 and Week 12 | Week 1, Week 4, Week 8 and Week 12 after treatment
  The DAS consists of the four domains hygiene, dressing, limb position and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Incidence of Adverse Events and Serious Adverse Events | Within 12 weeks of treatment
Incidence of Anti-drug Antibodies and Neutralizing Antibodies | Within 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Wan, Principal Investigator — Peking Union Medical College Hospital
Locations (24):
- China (24):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Henan University, Kaifeng, Henan
  - RenMin Hospital Of Wuhan University, Wuhan, Hubei
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - Qilu Hospital of Shandong University, Qingdao, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Rui Jin Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Fudan University HuaShan Hospital, Shanghai, Shanghai Municipality
  - Yangzhi Affiliated Rehabilitation Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi provincial people's Hospital, Taiyuan, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No